CLINICAL TRIAL: NCT05545527
Title: Neuroimaging Ancillary Study of the IV Iron RAPIDIRON Trial
Brief Title: Neuroimaging Ancillary Study
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Jawaharlal Nehru Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: U32401
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Iron Deficiency Anemia; Iron Deficiency Anemia of Pregnancy; Neurodevelopmental Disorder of Foetus; Iron Deficiency Anemia Treatment; Fetal Neurodevelopmental Disorder; Child Development
Keywords: India; Neuroimaging; Intravenous iron; MRI; Pediatrics
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; iron isomaltoside 1000; ferric derisomaltose; ferric sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- RAPIDIRON IV iron intervention arm 1: Maternal participants in this arm were given a single dose of an IV iron formulation - ferric carboxymaltose - during pregnancy as part of their participation in the parent RAPIDIRON Trial. Participants weighing 50kg and over received a single dose having 1000mg of iron, with others receiving a lower dose as determined by a formula used by the manufacturer (20mg iron/kg body weight). This was given between 14 and 17 weeks fetal gestational age.
  Interventions: Drug: Ferric carboxymaltose
- RAPIDIRON IV iron intervention arm 2: Maternal participants in this arm were given a single dose of an IV iron formulation - iron isomaltoside - during pregnancy as part of their participation in the parent RAPIDIRON Trial. Participants weighing 50kg and over received a single dose having 1000mg of iron, with others receiving a lower dose as determined by a formula used by the manufacturer (20mg iron/kg body weight). This was given between 14 and 17 weeks fetal gestational age.
  Interventions: Drug: Iron isomaltoside
- RAPIDIRON active comparator arm: Maternal participants in this arm of the RAPIDIRON Trial were given ferrous sulfate tablets with 60mg elemental iron each and instructed to take two per day (one in the morning and one at night) throughout their pregnancy.
  Interventions: Drug: Ferric Sulfate

INTERVENTIONS:
Drug: Ferric carboxymaltose — As part of the RAPIDIRON Trial, maternal participants randomized to intervention arm 1 were given a single dose of ferric carboxymaltose between 14 and 17 weeks of pregnancy.
  Groups: RAPIDIRON IV iron intervention arm 1
Drug: Iron isomaltoside — As part of the RAPIDIRON Trial, maternal participants randomized to intervention arm 2 were given a single dose of iron isomaltoside between 14 and 17 weeks of pregnancy.
  Other Names: Ferric derisomaltose
  Groups: RAPIDIRON IV iron intervention arm 2
Drug: Ferric Sulfate — As part of the RAPIDIRON Trial, maternal participants randomized to the active comparator arm were given 200 ferrous sulfate tablets immediately after randomization (~12 weeks of pregnancy). Participants were instructed to take two tablets a day, with each tablet containing 60mg elemental iron.
  Other Names: Ferric sulphate
  Groups: RAPIDIRON active comparator arm

SUMMARY:
As a follow-up to the RAPIDIRON Trial (NCT05358509), and in combination with the RAPIDIRON-KIDS Study (NCT05504863), this study will involve infants of RAPIDIRON Trial participants recruited at one site in Karnataka and is designed to implement a magnetic resonance imaging (MRI) protocol and incorporate neuroimaging measures. Implementation of this study will promote an understanding of the effects on fetal and neonatal brain development, including iron deposition in brain tissues, when a woman is treated for iron deficiency anemia (IDA) by either (a) providing her oral iron tablets and instructions for use; or (b) administering a single-dose IV iron infusion for the treatment of IDA during pregnancy.

DETAILED DESCRIPTION:
The hypothesis of this study is as follows:

* Reduced iron availability through fetal development impacts fundamental early neurodevelopmental processes, including neurogenesis of the hippocampus, amygdala, and other 'core' deep brain basal ganglia regions (e.g., globus pallidus); and myelination of the brain's white matter connecting these deep brain structures and higher-order cortical regions involved in motor, memory, and executive functioning.

The specific aims of this Neuroimaging Ancillary Study are:

* To determine impact of the IV iron intervention compared to oral iron on specific markers of brain development; and
* As a secondary analysis, to explore whether infant sex acts as a moderator of treatment on these specific brain development markers.

This study will recruit pregnant mothers currently participating in the parent RAPIDIRON Trial, who will be approached to give consent for themselves and their offspring for participation in this Neuroimaging Ancillary Study. Participation in this Ancillary Study will involve assessments at 32-35 weeks fetal gestational age, birth, 4 months, 12 months, and 24 months post-delivery. This will involve a fetal MRI and three post-birth MRIs conducted with the offspring to collect the main neuroimaging measures. In addition, we will collect various secondary offspring and maternal measures including child auditory brain response; maternal depression, anxiety, perceived stress, and empowerment; hair cortisol; and breastmilk micronutrient analysis.

Please see the protocol for additional details.

ELIGIBILITY:
Inclusion Criteria:

* For the maternal participant in the parent RAPIDIRON Trial - a pregnancy that has not gone beyond the period for obtaining a fetal MRI (by scanning the mother at 32-35 weeks fetal gestational age)
* An indication of the pregnant woman's intent to deliver in the study area and to reside there so as to be available not only to complete RAPIDIRON participation but also to allow her and her offspring to participate in ancillary study visits;
* Informed consent of the pregnant RAPIDIRON participant for her participation and that of her offspring in this ancillary trial; and
* Concurrent participation in the RAPIDIRON-KIDS follow-up study (NCT05504863).

Exclusion Criteria:

* If a fetal brain anomaly is found when the maternal participant undergoes an MRI at 32-35 weeks fetal gestational age, the dyad would be excluded from the ancillary study;
* If any of the following occur, this would result in dyad ineligibility for participation or continued participation in this ancillary study: maternal blood transfusion after enrollment, a pregnancy ending in stillbirth, neonatal death, diagnosis in the offspring of moderate to severe hypoxic-ischemic encephalopathy (or HIE), and/or blood transfusion to the offspring.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: For this ancillary study, only infants of randomized RAPIDIRON Trial (NCT05358509) participants recruited in Karnataka State will be eligible for participation.
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Fetal hippocampal volume | 32-35 weeks fetal gestational age
  Fetal hippocampus volume, measured via fetal MRI
Fetal diffusion parameters: fractional anisotropy (FA) | 32-35 weeks fetal gestational age
  Fetal white matter microstructure will be measured via FA at the posterior limb of internal capsule using fetal MRI
Fetal diffusion parameters: mean diffusivity | 32-35 weeks fetal gestational age
  Fetal white matter microstructure will be measured via MD at the posterior limb of internal capsule using fetal MRI

SECONDARY OUTCOMES:
Fetal sub-cortical gray matter structures | 32-35 weeks fetal gestational age
  Fetal sub-cortical gray matter structures in the brain using fetal MRI
Fetal white matter microstructure measures | 32-35 weeks fetal gestational age
  Additional fetal white matter microstructure measures using fetal MRI, including qualitative T2 MRI measures and NODDI metrics
Child hippocampal volume | 4 - 24 months of age
  Child hippocampal volume, measured via MRI
Child white matter volume | 4 - 24 months of age
  Child white matter volume, measured via MRI
Child white matter microstructure | 4 - 24 months of age
  Child white matter microstructure, including myelination, fiber coherence, and architecture, measured via MRI
Child white matter connectivity | 4 - 24 months of age
  Child white matter connectivity, measured via MRI
Child functional connectivity | 4 - 24 months of age
  Child functional connectivity, measured via MRI
Child cerebral metabolism | 4 - 24 months of age
  Child cerebral metabolism, including perfusion and spectroscopy, measured via MRI

OTHER OUTCOMES:
Child auditory brain response (ABR) results | Birth - 4 months of age
  Results on auditory brain response test
Hair cortisol results | Birth
  Results from hair cortisol testing
Maternal depression | Measured from 32-35 weeks fetal gestational age - 24 months offspring age
  Maternal depression, measured via the Edinburgh Post-Natal Depression Scale
Maternal anxiety | Measured from 32-35 weeks fetal gestational age - 24 months offspring age
  Maternal anxiety, measured via State-Trait Anxiety Inventory
Maternal Perceived Stress | Measured from 32-35 weeks fetal gestational age - 24 months offspring age
  Maternal Perceived Stress, measured via the Perceived Stress Scale (PSS-10)
Maternal Empowerment | Measured from 32-35 weeks fetal gestational age - 24 months offspring age
  Maternal empowerment, measured via the SWPER Global Survey
Breastmilk micronutrient analysis | 4 months offspring age
  Breastmilk micronutrient analysis, measured via maternal breastmilk samples
Maternal iron status | 32 - 35 weeks fetal gestational age
  Maternal iron status, measured via hemoglobin, ferritin and TSAT

CONTACTS AND LOCATIONS:
Overall Officials: Richard Derman, MD, MPH, Principal Investigator — Thomas Jefferson University
Locations (1):
- Jawaharlal Nehru Medical College, Belagavi, Karnataka, India